CLINICAL TRIAL: NCT05260684
Title: Comparative Effectiveness of Different Targeted Therapies for BRAF-mutated Unresectable/Metastatic Melanoma in the United States
Brief Title: Comparative Effectiveness of Targeted Therapies in BRAF Positive Metastatic Melanoma in the US
Acronym: OCEANMIST
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4221028; OCEANMIST (Other: Alias Study Number)
Record Dates: First submitted 2022-01-11; First posted 2022-03-02 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Melanoma
Keywords: BRAF-mutant; Metastatic melanoma
MeSH Terms: conditions — Melanoma | interventions — encorafenib; Drug Administration Routes; binimetinib; Vemurafenib; cobimetinib; dabrafenib; trametinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Encorafenib + binimetinib: Encorafenib 450 mg once a day (QD) Binimetinib 45 mg twice a day (BID)
  Interventions: Drug: Encorafenib; Drug: Binimetinib
- Vemurafenib + Cobimetinib: Vemurafenib 960 mg twice a day (BID) for 28 days of 28 day cycle Cobimetinib 60 mg once a day (QD) for 21 days of 28 day cycle
  Interventions: Drug: Vemurafenib; Drug: Cobimetinib
- Dabrafenib + trametinib: Dabrafenib 150 mg twice a day (BID) Trametinib 2 mg once a day (QD)
  Interventions: Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Encorafenib — 450 mg QD
  Other Names: Administration route: Oral
  Groups: Encorafenib + binimetinib
Drug: Binimetinib — 45 mg BID
  Other Names: Administration route: Oral
  Groups: Encorafenib + binimetinib
Drug: Vemurafenib — 960 mg BID for 28 days/cycle
  Other Names: Administration route: Oral
  Groups: Vemurafenib + Cobimetinib
Drug: Cobimetinib — 60 mg QD for 21 days/cycle
  Other Names: Administration route: Oral
  Groups: Vemurafenib + Cobimetinib
Drug: Dabrafenib — 150 mg BID
  Other Names: Administration route: Oral
  Groups: Dabrafenib + trametinib
Drug: Trametinib — 2 mg QD
  Other Names: Administration route: Oral
  Groups: Dabrafenib + trametinib

SUMMARY:
This study aims to compare real-world effectiveness of BRAF/MEK inhibitors in BRAF-mutant metastatic melanoma patients in the United States by line of therapy.

The Flatiron Health electronic health record (EHR) data from US cancer clinics will be used for this retrospective database analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with melanoma based on International Classification of Disease 9th and 10th Revisions (ICD-9: 172.x; ICD-10: C43x, D03x) and ≥2 visits on different days in the Flatiron database on or after January 1, 2011.
* Clinically confirmed diagnosis of melanoma with pathologic stages III or IV at initial diagnosis or earlier stage disease with a first locoregional or distant recurrence on or after January 1, 2011.
* Age ≥18 years at the time of advanced melanoma diagnosis.
* Evidence of ≥1 BRAF positive test result at any time based on laboratory or genetic analysis results.

Exclusion Criteria:

-• Patients with prior BRAF- or MEK-inhibitor therapy

• Patients with ECOG performance status ≥ 2 (at the time of randomization for patients from COLUMBUS, during the baseline period for patients in Flatiron EHR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be metastatic melanoma patients receiving targeted combination therapies derived from an anonymized Flatiron Health data combined with patient data from COLUMBUS trial data
Sampling Method: Non-Probability Sample
Enrollment: 716 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4221028

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of eligible participants with v-Raf murine sarcoma viral oncogene homolog B protein (BRAF)V-600 mutant melanoma who aged greater than or equal to 18 years at the time of initiating treatment with encorafenib plus binimetinib (ENCO+BINI) or dabrafenib plus trametinib (DAB+TRAM) or vemurafenib plus cobimetinib (VEM+COBI) was collected retrospectively.
Pre-assignment Details: Data sources: COLUMBUS trial from 30-Dec-2013-15-Sept-2020 [approximately 80.5 months] and Flatiron Health electronic health Records (EHR) real-world database (RWD) from duration of 09-Jan-2014-30-Sep-2021 [92.7 months]. Planned cohorts in this study: 1) ENCO+BINI, pooled across COLUMBUS and Flatiron EHR; 2) DAB+TRAM: from Flatiron EHR; 3) VEM+COBI: from Flatiron EHR. Available retrospective data was evaluated in this observational study from 17-Jan-2022-31-Dec-2023 (approximately 23.5 months).
Groups:
- Encorafenib+Binimetinib: Participants with BRAFV600-mutant metastatic melanoma, who were enrolled between 30-December 2013 to 15-September-2020 in phase 3 COLUMBUS trial and eligible participants from RWD cohort identified from Flatiron Health Database between 27-June-2018 to 30-September- 2021 and treated with Encorafenib 450 mg once daily (QD) and Binimetinib 45 mg twice daily (BID)(ENCO+BINI) were included.
- Dabrafenib+Trametinib: Eligible participants from RWD cohort with BRAFV600-mutant metastatic melanoma identified from Flatiron Health Database between 09-January-2014 to 30-September-2021 and treated with Dabrafenib 150 mg BID+ Trametinib 2 mg QD (DAB+TRAM) were included.
- Vemurafenib + Cobimetinib: Eligible participants from RWD cohort with BRAFV600-mutant metastatic melanoma identified from Flatiron Health Database between 10-November-2015 to 30-September-2021 and treated with Vemurafenib 960 mg BID+ Cobimetinib 60 mg QD (VEM+COBI) were included.
Period: Overall Study
Arm/Group | Encorafenib+Binimetinib | Dabrafenib+Trametinib | Vemurafenib + Cobimetinib
Started | 275 | 387 | 54
Completed | 275 | 387 | 54
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible participants whose data was retrieved and observed in the study.
Groups:
- Encorafenib+Binimetinib: Participants with BRAFV600-mutant metastatic melanoma, who were enrolled between 30-December 2013 to 15-September-2020 in phase 3 COLUMBUS trial and eligible participants from RWD cohort identified from Flatiron Health Database between 27-June-2018 to 30-September- 2021 and treated with Encorafenib 450 mg QD and Binimetinib 45 mg BID (ENCO+BINI) were included.
- Total: Total of all reporting groups
Arm/Group | Encorafenib+Binimetinib | Dabrafenib+Trametinib | Vemurafenib + Cobimetinib | Total
Number analyzed (Participants) | 275 | 387 | 54 | 716
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.5 (13.9) | 59.3 (13.5) | 56.4 (14.6) | 58.4 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 151 | 17 | 281
  Male | 162 | 236 | 37 | 435
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 253 | 353 | 48 | 654
  Non-white | 22 | 34 | 6 | 62

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: As per COLUMBUS trial, OS was defined as the time from the date of randomization to the date of death due to any cause; if death was not observed, participants were censored at the date of last contact or the data analysis cut-off date, whichever occurred first. As per Flatiron EHR, OS was defined as the time from the index date to the date of death; participants without a date of death were censored at their last known activity date or the end of the follow-up period, whichever occurred first. Index date in each treatment group was defined as the date of treatment initiation. Kaplan-Meier analyses was used for analysis.
Time Frame: COLUMBUS: From date of randomization until death or censoring (approx 80.5 months); Flatiron: From index date until death due or censoring or end of follow-up period (92.7 months)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dabrafenib+Trametinib | Vemurafenib + Cobimetinib | Encorafenib+Binimetinib
Number analyzed (Participants) | 387 | 54 | 275
Months | 16.1 [13.7 to 18.7] | 25.0 [17.0 to NA] — To estimate an upper limit of 95% confidence limit (CI), enough follow-up and events were required after the median OS reached. But beyond median OS, participants at risk and events were insufficient. Hence, upper limit of 95% CI could not be estimated. | 30.0 [24.4 to 37.6]
Statistical Analysis 1: Comparison: Dabrafenib+Trametinib vs Encorafenib+Binimetinib; Statistical analysis data is presented for Dabrafenib+Trametinib relative to Encorafenib+Binimetinib (reference); Test type: Other; p = 0.02, Wald Chi- Square Statistic; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [1.05 to 1.65] — HR was estimated using multivariable Cox proportional hazard models
Statistical Analysis 2: Comparison: Vemurafenib + Cobimetinib vs Encorafenib+Binimetinib; Statistical analysis data is presented for Vemurafenib + Cobimetinib relative to Encorafenib+Binimetinib (reference); Test type: Other; p = 0.47, Wald Chi- Square Statistic; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.76 to 1.79] — HR was estimated using multivariable Cox proportional hazard models

2. Other Pre Specified Outcome: Progression Free Survival (PFS)
Description: COLUMBUS:PFS=time from the date of randomization to the date of the first documented disease progression (PD) or death due to any cause, whichever occurred first; PD:at least 20 percentage (%) increase in the sum of diameter of all measured target lesions, reference to the smallest sum of diameter of all target lesions recorded at or after baseline. In addition, increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimiter square (mm2) or the appearance of 1 or more new lesion, if a participant did not have an event at the analysis cut-off date, PFS was censored at the date of the last adequate tumour assessment. Flatiron:PFS=time from the index date to either the date of first PD event or death in the absence of progression; participants without PD or death were censored at the last date the participant could have been assessed for progression or the data analysis cut-off date, whichever occurred first. Index date was =the date of treatment initiation.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dabrafenib+Trametinib | Vemurafenib + Cobimetinib | Encorafenib+Binimetinib
Number analyzed (Participants) | 387 | 54 | 275
Months | 7.4 [6.3 to 8.4] | 7.9 [5.5 to 24.4] | 14.1 [11.4 to 17.7]
Statistical Analysis 1: Comparison: Dabrafenib+Trametinib vs Encorafenib+Binimetinib; Statistical analysis data is presented for Dabrafenib+Trametinib relative to Encorafenib+Binimetinib (reference); Test type: Other; p < 0.001, Wald Chi- Square Statistic; Hazard Ratio (HR) = 1.49, 95% CI 2-sided [1.20 to 1.87] — HR was estimated using multivariable Cox proportional hazard models
Statistical Analysis 2: Comparison: Vemurafenib + Cobimetinib vs Encorafenib+Binimetinib; Statistical analysis data is presented for Vemurafenib + Cobimetinib relative to Encorafenib+Binimetinib (reference); Test type: Other; p = 0.40, Wald Chi- Square Statistic; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.79 to 1.82] — HR was estimated using multivariable Cox proportional hazard models

ADVERSE EVENTS:
Time Frame: All-cause mortality: COLUMBUS trial from 30-December-2013 to 15-September-2020 [approximately 80.5 months] and Flatiron EHR RWD from duration of 09-January-2014 to 30-September-2021 [92.7 months]; For adverse events it was not applicable as adverse event data was not planned to be collected.
Description: This study is retrospective, it involves data that exist as structured data by the time of study start. The minimum criteria for reporting an adverse event (AE) (i.e., identifiable participant, identifiable reporter, a suspect product, and event) cannot be met. Hence, adverse events were not planned to be collected and are not reported.
Arm/Group | Encorafenib+Binimetinib | Dabrafenib+Trametinib | Vemurafenib + Cobimetinib
All-Cause Mortality (participants affected / at risk) | 159/275 | 259/387 | 30/54
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT05260684/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT05260684/SAP_001.pdf